CLINICAL TRIAL: NCT04595409
Title: A Randomised, Double-blind, Parallel-group, Phase 3 Study to Compare the Efficacy, Safety, and Immunogenicity of the Proposed Biosimilar Ustekinumab FYB202 to Stelara® in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Double-blind Study to Compare the Efficacy, Safety, and Immunogenicity of the Proposed Biosimilar Ustekinumab FYB202 to Stelara® in Patients With Moderate-to-Severe Plaque Psoriasis
Acronym: VESPUCCI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bioeq GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FYB202-03-01
Record Dates: First submitted 2020-10-14; First posted 2020-10-20 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Ustekinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FYB202 (Proposed ustekinumab biosimilar) (Experimental): Patients will receive subcutaneous injections of FYB202 as detailed in the protocol.
  Interventions: Drug: FYB202 (Proposed ustekinumab biosimilar)
- Stelara® (Ustekinumab) (Active Comparator): Patients will receive subcutaneous injections of Stelara® as detailed in the protocol.
  Interventions: Drug: Stelara® (Ustekinumab)

INTERVENTIONS:
Drug: FYB202 (Proposed ustekinumab biosimilar) — Patients will receive 1 subcutaneous (SC) injection of FYB202 at week 0 and week 4, followed by 1 SC injection every 12 weeks thereafter for the next 3 consecutive doses.
  Arms: FYB202 (Proposed ustekinumab biosimilar)
Drug: Stelara® (Ustekinumab) — Patients will receive 1 subcutaneous (SC) injection of Stelara® at week 0 and week 4, followed by 1 SC injection every 12 weeks thereafter for the next 3 consecutive doses.
  Arms: Stelara® (Ustekinumab)

SUMMARY:
This is a randomized, double-blind, multicenter study to evaluate the efficacy, safety, and immunogenicity of FYB202 compared to Stelara® in patients with Moderate-to-Severe Plaque Psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who provided written informed consent and who are able to complete study procedures.
2. Patients who are at least 18 years of age at time of screening.
3. Patients with PASI score of at least 12 at screening and at baseline.
4. Patients with involved body surface area of at least 10% at screening and at baseline.
5. Patients with a Physician's Global Assessment (PGA) score of at least 3 at screening and at baseline by means of a 5-point scoring scale.
6. Patients who are candidates for systemic therapy or phototherapy.
7. Previous failure, inadequate response in the opinion of the investigator, intolerance, or contraindication to at least 1 conventional antipsoriatic systemic therapy.
8. For female patients (except those at least 2 years postmenopausal or surgically sterilised): a negative serum pregnancy test at screening and at baseline.
9. Female patients of childbearing potential with a fertile male sexual partner must use adequate contraception from screening until 4 months after the last dose of study intervention. Adequate contraception is defined as using hormonal contraceptives or an intrauterine device (IUD), combined with at least one of the following forms of contraception: a diaphragm, cervical cap, or a condom. Total abstinence from heterosexual activity, in accordance with the lifestyle of the patient, is acceptable. Female patients must not donate ova starting at screening and throughout the clinical study period and for 4 months after study intervention administration.
10. Male patients who are sexually active with women of childbearing potential must agree they will use adequate contraception if not surgically sterilised and will not donate sperm from the time of screening until 6 months after the last dose of study intervention. Adequate contraception for the male patient and his female partner of childbearing potential is defined as using hormonal contraceptives or an IUD combined with at least one of the following forms of contraception: a diaphragm, cervical cap, or a condom. Total abstinence from heterosexual activity, in accordance with the lifestyle of the patient, is acceptable.

Exclusion Criteria:

1. Patients diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, medication-induced psoriasis, any other skin disease, or other systemic inflammatory autoimmune disorder at the time of the screening and baseline visits that would interfere with evaluations of the effect of study intervention on psoriasis.
2. Patients who have received any topical psoriasis treatment including corticosteroids.
3. Patients who have received the following treatments for psoriasis:

   1. PUVA phototherapy and/or ultraviolet B phototherapy and/or laser therapy
   2. Non-biologic psoriasis systemic therapies, tofacitinib, or apremilast
   3. Adalimumab
   4. Etanercept or secukinumab
   5. Infliximab, brodalumab, certolizumab pegol, ixekizumab, golimumab, or alefacept
4. Patients taking drugs that may cause new onset or exacerbation of psoriasis
5. Patients who have received ustekinumab or any biologics directly targeting interleukin (IL) 12 or IL 23.
6. Patients with active infection or history of infections as follows:

   1. Any active infection for which systemic anti-infectives were used within 4 weeks prior to randomisation
   2. A serious infection, defined as requiring hospitalisation or intravenous anti-infectives, within 8 weeks prior to randomisation
   3. Evidence of any clinically relevant bacterial, viral, fungal, or parasitic infection
   4. Recurrent or chronic infections or other active infection that, in the opinion of the investigator, might cause this study to be detrimental to the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 392 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Percent improvement in Psoriasis Area and Severity Index (PASI) score | Week 12

SECONDARY OUTCOMES:
Percent improvement in PASI score | Through study completion, approximately 1 year
Raw PASI score | Through study completion, approximately 1 year
Proportion of patients with PASI 75 and PASI 90 | Through study completion, approximately 1 year
Change per Physician's Global Assessment (PGA) | Through study completion, approximately 1 year
Improvement of Dermatology Life Quality Index (DLQI) total score | Through study completion, approximately 1 year
Itching Visual Analogue Scale | Through study completion, approximately 1 year
Relative frequency, nature, and severity of adverse events (AEs) and serious adverse events (SAEs) | Through study completion, approximately 1 year
Serum trough levels of ustekinumab | Through study completion, approximately 1 year
Number of patients with antibodies to ustekinumab | Through study completion, approximately 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Study Official, Study Director — Bioeq GmbH
Locations (16):
- Estonia (2):
  - Research Site, Tallinn
  - Research Site, Tartu
- Research Site, Tbilisi, Georgia
- Poland (8):
  - Research Site, Bialystok
  - Research Site, Gdansk
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Olsztyn
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Ukraine (5):
  - Research Site, Dnipro
  - Research Site, Kharkiv
  - Research Site, Kyiv
  - Research Site, Rivne
  - Research Site, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Papp K, Balser S, Nopora K, Rewerski P, Freudensprung B, Trieb M. A Randomised, Double-Blind Trial to Compare the Efficacy, Safety, and Immunogenicity of the Biosimilar Ustekinumab FYB202 with Reference Ustekinumab in Patients with Moderate-to-Severe Plaque Psoriasis. Adv Ther. 2025 May;42(5):2135-2149. doi: 10.1007/s12325-025-03138-2. Epub 2025 Mar 6. PMID 40048101